# **Study Protocol**

**Official title**: Effectiveness Study of Two Types of Intervention for People in Couple Who Have Difficulties With Their Gambling Habits or Alcohol/Drug Use

NCT number: NCT05833503

**Document date**: 2024-04-06

Principal Investigator: Joël Tremblay (418) 659-2170, #2820

This project has been approved by UQTR's research ethics committee (CERPPE-21-01-10.01) and the research ethics committee of the Centre intégré de santé et de services sociaux de Chaudière-Appalaches (MP-23-2022-894).

Document date: 2024-04-06.

### Random distribution research design

The efficacy study, using a longitudinal mixed methods approach, is conducted with a randomization process (n=100 couples) whereby participants are assigned to one of two treatment groups: a) an experimental group involving couple counselling (n = 50), and b) a control group involving individual counselling (n = 50). After the evaluation interview, the research officer applies randomization to ensure that each participant is randomly assigned to one of the two interventions. The method used is urn randomization (Wei and Lachin, 1988), combined with stratification for covariates thought to influence treatment outcome (Hedden, Woolson and Malcolm, 2006).

# Stratification criteria (covariates) for randomization

- The Gambler presents significant gambling problems (PGSI  $\geq$  8) as well as alcohol or other psychoactive substance use (ASSIST  $\geq$  27).
- The Gambler has a gambling disorder (PGSI  $\geq$  8).
- The Gambler is cisgender female.
- The Gambler has a gender identity other than cisgender male or cisgender female.
- The Partner has a moderate problem with substance use (score between 11-26 on ASSIST for alcohol, 4-26 for other substances) or gambling (score between 3-7 on PGSI).
- Presence of significant mental health problems, stabilized in either the Gambler OR their Partner over the past year:
  - Current mental well-being according to *The World Health Organization-Five Well-Being Index* (WHO-5) score ≤ 50 (WHO, 1999).
  - o Significant psychological distress, 85th percentile on the *Psychological Distress Index of the Quebec Health Survey* IDPESQ-14 score ≥ 31 for women or ≥ 27 for men (Préville, Boyer, Potvin, Perreault, & Légaré, 1992).
  - O Severity of borderline personality disorder on the *Borderline Symptom List (BSL-23)* score  $\geq 0.8$  (Bohus et al., 2009).
  - o Indicator of the presence of another personality disorder, *Standardised Assessment of Personality Abbreviated Scale (SAPAS)* score ≥ 4 (Moran, Leese, Lee, Walters, Thornicroft, & Mann, 2003) Adaptation by Ferland and Blanchette-Martin (2010) and *The Narcissistic Grandiosity Scale (NGS)* score ≥ 6 (Rosenthal et al., 2020).
- All other couples consisting of non-heterosexual partners.

**Participants** 

Participants will be recruited from the specialized addiction services (also called addiction

rehabilitation centers) of ten Centre intégré de santé et de services sociaux/Centre intégré universitaire de santé et de services sociaux, namely those of the Capitale-Nationale, Chaudière-

Appalaches, Centre-sud de l'Île de Montréal, Montérégie Ouest, Lanaudière, Laurentides, Eastern

Townships, Saguenay-Lac-St-Jean, Laval and Mauricie-Centre-du-Québec regions. These

establishments serve more than 80% of the Quebec population.

Selection criteria

Inclusion Criteria:

• The Gambler may have a gambling or substance use problem at the beginning of treatment

AND is accepted for treatment by addiction rehabilitation centers (CRDs).

• The Gambler has engaged in gambling or substance use behaviors in the past three months

(Time Line Follow-Back).

The Partner may or may not engage in gambling, consume alcohol or other substances of

abuse.

• Living in couple for at least six months OR report being in a significant relationship for at

least two years.

Exclusion Criteria:

• The Gambler has been completely abstinent from any gambling or substance use problem

for the past three months.

• The Gambler received treatment for gambling disorder or substance abuse disorder during

the last six months (excluding Gamblers Anonymous, Alcoholics Anonymous or Narcotics

Anonymous).

• Low level of marital commitment between the couple in the past 2 weeks indicating a high

risk of short-term separation (Marital Status Inventory, score  $\geq 9$ )

• Presence of serious acts of violence committed within the past year endangering the safety

or life of one of the spouses (*Modified Conflict Tactics Scales*: Answer YES to any question

from Q27-33) OR use of services for victims of domestic violence in the past year.

3

Document date: 2024-04-06.

• Presence of an active mental health disorder in either partner hindering therapeutic participation, such as a psychotic disorder OR a suicide attempt in the last 30 days (Psychological Scale of the Addiction Severity Index) OR severe borderline personality disorder (BSL-23 ≥2.8) OR excessively extreme antisocial behaviors (Conduct Disorder Scale from the GAIN ≥ 9).

# Recruitment strategies

Generally, practitioners propose the study to users following routine admission evaluations in the participating centres. Individuals interested in participating sign a form authorizing a research officer to contact them. A research assistant then reaches out to gambler who have accepted to be contacted and explains the research project in more detail to the person and the spouse; a first meeting with the couple is also set. During the meeting, once the questionnaires have been completed, randomization is carried out and the couple told about the intervention method to which they have been randomly assigned. In all cases, spouses are informed that they can get support from the entourage program (individual or group) offered in all participating centres.

In light of each centre's usual service request process, the recruitment strategy has been adapted to the realities of each one so as to facilitate referrals.

A poster describing the research project has also been produced and put up in the waiting rooms of all participating centres. A flyer based on the poster has also been made so clinicians can give out information about the study to anyone interested.

# Intervention requirements

Document date: 2024-04-06.

- A) Experimental group: Integrative Couple Treatment for Addiction (ICT-A) Inspired by the "Alcohol Behavior Couple Therapy" from Epstein & McCrady, the ICT-A will be offered over 12 to 16 sessions of 90 minutes. Typically, approximately the first half of each session is dedicated to GD/SUD problems,in a predominantly cognitive behavioral model. In the second part of each session, the clinician will help the couple to improve their communication,to reduce the reinforcements (non-voluntary) of the behaviors of GD/SUD and to increase marital pleasure situations incompatible with the use of GD/SUD.Particular attention will also be paid to feelings of betrayal and interpersonal attacks to restore trust. Plus, they will received a sefl-care guide.
- B) Control group: Individual treatment as usually offered

  The usual treatment control group will receive individual treatment as already offered by
  the specialized centres in addiction.

  For the person with GD/SUD, this treatment consists of 12 to 16 individual cognitive-

For the person with GD/SUD, this treatment consists of 12 to 16 individual cognitivebehavioral sessions of 60 minutes. In general, the intervention aims to secure financial assets, awareness of erroneous thoughts and improvement of alternative skills to gambling in order to meet the normal demands of psychic and relational life. People undergoing this intervention will receive a self-care guide.

As for the partners randomized in this intervention, they will receive the services that are usually offered to members of the entourage of a person with GD/SUD. In groups or individually, these services are generally aimed at improving the partner's well-being and relationship with their spouse, which includes information about GD/SUD and the recovery process.

#### Research process

Following admission to treatment, an 18-month longitudinal follow-up will document the effects of the intervention and the maintenance of gains over time. The research assessments will therefore take place on four occasions, at intake, 6-, 12 and 18-months post-admission.

The initial meeting takes place before therapy sessions begin; the second is held about six months after, and the third about 12 months after onset of therapy. A last meeting is held 18 months after the start of participation in the project. During the sessions, participants complete a series of questionnaires on lifestyle habits, personal state, and conjugal life.

Following the first meeting with the research officer, the latter contacts the couple or referring practitioner again (depending on the outcome of the evaluation meeting) within 24 hours to confirm or reject the couple's participation in the project. If a couple is chosen for the research project, the referring practitioner contacts them to inform them of treatment plan to which they are being referred and to schedule a meeting. If the couple has not been chosen (exclusion criteria), the research assistant who conducted the admission interview contacts the couple to inform them of the decision. In this case, the referring practitioner is also notified of the meeting's outcome so the player and his or her spouse can benefit from the services which they could normally obtain in the centre where the initial request for help was made.

If a couple is assigned to couple therapy, the research officer sends a summary of the evaluation findings to the clinician to help him or her better understand the couple's situation and preclude having to ask for the same information a second time. Also, at the beginning of each treatment meeting, both members of the couple complete a few brief 15-minute questionnaires on lifestyle habits and certain aspects of conjugal life.

The clinician films the couple sessions for supervision meetings with study researchers (a session every month), so the therapist can intervene as effectively as possible to help the couple.

The monetary compensation offered will be \$275 per couple, offered in the form of gift cards to a local mall (\$50 at the first intake meeting, \$75 at the three meetings 6, 12 and 18 months post-intake). Since participants are expected to attend four research meetings over a year and a half, as well as 12 to 16 treatment meetings, we believe that the \$275 per couple compensation is commensurate with the effort required.

# Training for clinicians

The research team organized three day of training sessions for participating clinicians. During these sessions, the clinical model was presented, including training on the use of functional analysis for gambling situations and situations presenting risks of relapse, basic principles of couple therapy, strategies to improve communication, quality of negotiation, reduction of behaviours that reinforce gambling habits, and bolstering behaviours incompatible with gambling.

# Treatment quality control

At the end of each interview (individual treatment or couple treatment), the clinician clinicians complete a checklist rating the importance of each theme during the encounter (scale of 0 to 10 where 0 = not at all, 10 = extremely).

Supervision sessions are also a way to verify the quality of application of the intervention model evaluated.

6